CLINICAL TRIAL: NCT00900861
Title: Asthma Control and Clinical Practice in Hungary 2009
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MCMD, AstraZeneca
Other Study IDs: NIS-RHU-DUM-2009/1
Record Dates: First submitted 2009-05-12; First posted 2009-05-13 (Estimated); Last update posted 2009-12-04 (Estimated); Status verified 2009-12

CONDITIONS: Asthma Control Level
Keywords: asthma control level; visual analogue scale

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Asthmatic patients above 18 y, treated with ICS or bronchodilators

SUMMARY:
A prospective study led amongst pulmonologists. Patients asthma control level will be evaluated based on GINA guideline criteria. HRQoL measured by Visual analogue scale. Clinical practice: non controlled patients therapy assessed.

ELIGIBILITY:
Inclusion Criteria:

* Asthma patients treated with ICS or bronchodilators

Exclusion Criteria:

* COPD
* pulmonary cancer
* pulmonary tuberculosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Pulmonology outpatient clinics
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2009-04; Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Asthma control level | 3 times

SECONDARY OUTCOMES:
Visual Analogue Scale | 3 times
Routine Therapeutical habits in control maintenance | 3 times

CONTACTS AND LOCATIONS:
Overall Officials: Zoltan Bartfai, MD PhD, Principal Investigator — Semmelweis University Budapest Pulmonology Clinic; Lilla Szabo, Study Chair — AstraZeneca Hungary; Eva Gulyas, Study Director — AstraZeneca Hungary
Locations (75):
- Hungary (75):
  - Research Site, Aszód
  - Research Site, Baja
  - Research Site, Baktalórántháza
  - Research Site, Balassagyarmat
  - Research Site, Bácsalmás
  - Research Site, Berettyóújfalu
  - Research Site, Békés
  - Research Site, Békéscsaba
  - Research Site, Bonyhád
  - Research Site, Cegléd
  - Research Site, Celldömölk
  - Research Site, Csorna
  - Research Site, Dabas
  - Research Site, Debrecen
  - Research Site, Dombóvár
  - Research Site, Dunaharaszti
  - Research Site, Dunaújváros
  - Research Site, Dunavecse
  - Research Site, Edelény
  - Research Site, Eger
  - Research Site, Encs
  - Research Site, Esztergom
  - Research Site, Érd
  - Research Site, Gávavencsellő
  - Research Site, Gödöllő
  - Research Site, Győr
  - Research Site, Győrújbarát
  - Research Site, Gyungyos
  - Research Site, Hajdúnánás
  - Research Site, Hatvan
  - Research Site, Ikrény
  - Research Site, Jászberény
  - Research Site, Kaposvár
  - Research Site, Kapuvár
  - Research Site, Kazincbarcika
  - Research Site, Keszthely
  - Research Site, Kisbér
  - Research Site, Kiskőrös
  - Research Site, Kiskunhalas
  - Research Site, Kistelek
  - Research Site, Kisvárda
  - Research Site, Mátészalka
  - Research Site, Mezőkövesd
  - Research Site, Miskolc
  - Research Site, Monor
  - Research Site, Mosonmagyaróvár
  - Research Site, Mór
  - Research Site, Nagyatád
  - Research Site, Nagykőrös
  - Research Site, Nyírbátor
  - Research Site, Nyíregyháza
  - Research Site, Orosháza
  - Research Site, Ózd
  - Research Site, Pápa
  - Research Site, Pásztó
  - Research Site, Pécs
  - Research Site, Salgótarján
  - Research Site, Sárbogárd
  - Research Site, Sárvár
  - Research Site, Siófok
  - Research Site, Szarvas
  - Research Site, Százhalombatta
  - Research Site, Szeged
  - Research Site, Szentendre
  - Research Site, Szerencs
  - Research Site, Szécsény
  - Research Site, Székesfehérvár
  - Research Site, Szolnok
  - Research Site, Tapolca
  - Research Site, Tata
  - Research Site, Tiszalök
  - Research Site, Tiszaújváros
  - Research Site, Törökbálint
  - Research Site, Vác
  - Research Site, Vásárosnamény